CLINICAL TRIAL: NCT01546610
Title: Effect of Rheumatoid Foot Insole
Brief Title: Rheumatoid Foot Insole
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Emilia Moreira, PT, Effect of rheumatoid foot insole, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1348/09
Record Dates: First submitted 2012-03-02; First posted 2012-03-07 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid foot; foot pain; insoles; foot function; electronic baropodometer; plantar pressure; gait analysis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intervention foot orthoses (Experimental): Ethyl vinyl acetate (EVA) insole with medial arch support and bar retrocapital
  Interventions: Other: insoles intervention
- placebo insole (Placebo Comparator): Foot orthose with support retrocapital and support of medial arch insole intervention
  Interventions: Other: placebo insole

INTERVENTIONS:
Other: insoles intervention — EVA insole with arch support and bar retrocapital
  Other Names: Interventional group
  Arms: intervention foot orthoses
Other: placebo insole — EVA insole flat
  Other Names: control group
  Arms: placebo insole

SUMMARY:
The present study aims to evaluate the effect of insoles for foot arthritis.

DETAILED DESCRIPTION:
A randomized, controlled, double-blind, prospective trial being conducted involving 80 patients with rheumatoid arthritis, according to American College of Rheumatology (ACR) criteria, and foot pain, selected from outpatient clinics - Federal University of Sao Paulo (UNIFESP).

Patients will be randomized in to two groups: experimental (40) and control (40).

The experimental group will use ethyl-vinyl acetate (EVA) foot orthoses, with support retrocapital and support of medial arch (insole intervention). The control group will use the same material flat insole (insole placebo).

ELIGIBILITY:
Inclusion Criteria:

* Patients with established diagnosis RA according to criteria of the American College of Rheumatology (ACR) functional classes I, II and III
* Foot pain with VAS between 3 - 8 cm for walking
* Age 18-65 years
* Basic medication stable for at least three months
* Not made infiltrations in feet and ankles in the last three months and not during the study
* Agreed to participate and signed term of informed consent

Exclusion Criteria:

* Other musculoskeletal disorders in symptomatic lower limbs
* Diseases of the central and peripheral nervous system
* Decompensated diabetes mellitus
* No walking
* Rigid deformities in the feet
* Use of insoles in the last three months
* Surgery scheduled in the next 12 months
* Allergy to the material
* Mental deficiency

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale of pain in feet during walking (VAS) | 12 months
  Assessing pain in the feet during walking through a visual analog scale from 0 to 10 centimeter (cm)

SECONDARY OUTCOMES:
Foot Function Index (FFI) | 12 months
  Function of the foot
Foot Health Status Questionnaire (FHSQ-Br) | 12 months
  Foot Health Status
Health Assessmente Questionnaire (HAQ) | 12 months
  Functional capacity assessed by HAQ in rheumatoid arthritis
Visual analog scale of pain in feet at rest (VAS) | 12 months
  Assessing pain in the feet at rest through a visual analog scale from 0 to 10
6-MINUTE WALK TEST | 12 months
  Assess functional capacity
Shorth Form-36 (SF-36) | 12 months
  Quality of life by SF-36
LIKERT SCALE | 12 months
  Likert scale by patients
TESTS BAROPODOMETRIC | 12 months
  Evaluates charge distribution in the feet and gait variables
TIME USE OF INSOLE | 12 months
  Control the use of time insole

CONTACTS AND LOCATIONS:
Overall Officials: EMILIA MOREIRA, PT, Principal Investigator — Federal University of São Paulo; ANAMARIA PT JONES, PHD, Study Director — Federal University of São Paulo; JAMIL NATOUR, PHD, Study Chair — Division of Rheumatology, Federal University of Sao Paulo
Locations (1):
- Emilia Moreira, São Paulo, São Paulo, Brazil